CLINICAL TRIAL: NCT02640274
Title: Self-management Behaviour After an Individual Nurse-led Counselling Programme for Patients Early Discharged After Myocardial Infarction: A Randomised Controlled Trial.
Brief Title: Individual Nurse-led Counselling Programme for Patients Early Discharged After Myocardial Infarction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013/1568/REK
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-10

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Myocardial Infarction
Keywords: Practise Patterns, Nurses'; Directive Counseling; Self Care
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Myocardial Infarction

ARMS (2):
- Intervention group (Experimental): The intervention is an individual nurse-led counselling programme in addition to usual care.
  Interventions: Behavioral: Nurse-led counselling programme; Other: Usual care
- Control group (Other): usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Nurse-led counselling programme — The intervention is an individual nurse-led counselling programme in addition to usual care. The intervention includes 3 outpatient clinic visits (at weeks 2, 14 and 26) and two telephone calls (at weeks 4 and 16) by a cardiovascular nurse during the first 6 months early discharged. The counselling focuses on cardiac risk reduction behaviour based on guidelines issued by European Society of Cardiology and self-management support.
  Arms: Intervention group
Other: Usual care

SUMMARY:
The European guidelines of cardiovascular disease prevention recommend treatment modalities, such as lifestyle changes in order to minimize the risk of further cardiac event after a myocardial infarction (MI). However, a considerable gap exists between guidelines and their implementation in clinical practise. Further, less is known about the impact of different interventions on patient's knowledge, skills and confidence necessary for self-management after MI.

Aim: To evaluate and compare the short- and long-term effects of an individual nurse-led counselling programme together with usual care for patients early discharged after MI on self-management behaviour.

ELIGIBILITY:
Inclusion Criteria:Patients with documented evidence of myocardial infarction during hospitalisation will be considered for inclusion.

* patients over 18 years old
* living at home in the local hospital area after hospital discharge
* able to receive telephone calls, fill in questionnaire and communicate in Norwegian.

Exclusion Criteria:

* cognitive impaired/dementia
* planning for coronary artery bypass graft surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-11; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Changes in self-management | from baseline to 6 and 12 months of follow-up
  Patient activation measure (PAM) consists of 13 items. The questionnaire assesses the patients' knowledge, skill and confidence for managing ones' own health care.

SECONDARY OUTCOMES:
changes in health behaviour | from baseline to 6 and 12 months of follow-up
  The SmartDiet questionnaire consists of 21 questions registering average use of certain group of food and lifestyle. The questions about physical activity is a questionnaire about frequency, duration and intensity of physical activities.

CONTACTS AND LOCATIONS:
Overall Officials: Liv Heidi Skotnes, phd, Principal Investigator — Leangen Hospital HNT
Locations (1):
- Medical Clinic, Namsos, Namsos, Norway